CLINICAL TRIAL: NCT03844893
Title: Macrophage Programing in Acute Lung Injury
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National Jewish Health (Other)
Responsible Party: Sponsor
Other Study IDs: HS-3076
Record Dates: First submitted 2019-02-12; First posted 2019-02-19 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-02

CONDITIONS: Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Mini bal — Mini-BAL is a minimally invasive technique frequently used in the investigator's local intensive care units (ICUs) to obtain alveolar fluid samples from mechanically ventilated patients. This is typically done for microbial analysis.

SUMMARY:
The histologic hallmarks of lung inflammation and in the extreme, acute respiratory distress syndrome (ARDS), include intense accumulation of inflammatory cells in the airspaces and interstitium, injury to alveolar epithelial and endothelial cells, loss of epithelial-capillary integrity and accumulation of edema fluid in the interstitium and airspaces. Accordingly, for alveolar repair to occur inflammation must be halted, debris and inflammatory cells removed, injured tissue cells replaced, and capillary barrier function re-established. Macrophages are key players in all of these. Here the investigators hypothesize that resident alveolar macrophages and recruited macrophages serve completely different functions, acting independently (i.e. division of labor) yet cooperatively (synergism).

ELIGIBILITY:
Inclusion Criteria:

1. Written, informed consent (by surrogate if unconscious or if altered mental status)
2. Admission to a Medical Intensive care unit
3. Orally/nasally intubated, evaluable within 24 h of intubation or onset of ARDS
4. Expected to remain mechanically ventilated for at least 48 h after the first study procedure.

Exclusion Criteria:

1. Treatment with immunosuppressants in the prior 3 months (antineoplastic agents, tumor necrosis factor alpha antagonists, cyclosporine, methotrexate, azathioprine, or mycophenolate. Treatment with glucocorticoids for septic shock is acceptable).
2. History of solid organ or bone marrow transplantation
3. History of chronic lung disease (e.g. COPD, pulmonary fibrosis, cystic fibrosis)
4. Human immunodeficiency virus positivity
5. Severe or massive hemoptysis
6. At significant risk for bleeding (INR > 3 or PTT > 3x normal)
7. Presence of an advanced directive to withhold life-sustaining treatment
8. Morbid state or expected to survive less than 14 days because of an advanced co-morbid medical condition;
9. Pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The population to be studied are patients identified to have ARDS, admitted to the intensive care unit, and placed on a mechanical ventilator. The MICU at National Jewish-St Joseph Hospital will be the primary site for enrollment. Control subjects will be individuals on mechanical ventilation for non-pulmonary reasons (i.e. following surgery, sepsis without lung involvement). A total of 56 subjects will be enrolled. As described below (in Research Methods and Enrollment) a 2:1 ratio of ARDS to control subjects will be targeted.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Estimated)
Dates: Start 2019-10 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Evaluation and roles of macrophages during ARDS | 10 days
  Evaluation of resident alveolar macrophages will be distinguished with flow cytometry and enumerated
Evaluation and roles of macrophages during ARDS | 10 days
  Evaluation of recruited alveolar macrophages will be isolated using FACS and subjected to RNA sequencing. Pro-inflammatory and pro-reparative modules will be assessed in the data set expression of transcription factors reported to drive macrophage polarization (HIF-1α, NF-kB, STAT-1, STAT-3, STAT-6, PPARγ, PU.1) will be assessed.